CLINICAL TRIAL: NCT03525626
Title: Online Mindfulness-based Tic Reduction: Development and Testing (Phase One)
Brief Title: Online Mindfulness-based Tic Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bowdoin College (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Hannah Reese, Assistant Professor, Bowdoin College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017-37
Record Dates: First submitted 2018-04-24; First posted 2018-05-15 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Tourette Syndrome; Tic Disorders
Keywords: Tic Disorders; Mindfulness; Meditation; Online; Internet-based; Treatment
MeSH Terms: conditions — Tourette Syndrome; Tic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Online Mindfulness-based Tic Reduction (Experimental)
  Interventions: Behavioral: Online Mindfulness-based Tic Reduction

INTERVENTIONS:
Behavioral: Online Mindfulness-based Tic Reduction — 8-week online group mindfulness-based intervention for tics

SUMMARY:
Tourette Syndrome (TS) and Persistent Tic Disorder (PTD) are chronic and potentially disabling neurobiological conditions. Although a range of pharmacological and psychosocial treatments exists, a significant number of individuals either do not respond to the current treatments, find them unacceptable, or cannot access them. Thus, it is essential that researchers continue to pursue novel treatment approaches that can also be easily disseminated to those in need.

Initial pilot data suggest that a mindfulness-based intervention may be beneficial for adults with tic disorders. In the present study, the researchers aim to further develop this mindfulness-based intervention, adapt it to be delivered online and pilot test the intervention with a small group of participants. The data from this pilot test will inform a subsequent randomized controlled trial comparing online mindfulness-based tic reduction to online psychoeducation, relaxation, and supportive therapy.

The specific aim is to determine the feasibility and acceptability of Online Mindfulness-based Tic Reduction in 6 adults with TS or PTD.

The researchers hypothesize that Online Mindfulness-based Tic Reduction will be feasible and acceptable to adults with tic disorders as measured by participant satisfaction, qualitative participant feedback, home practice compliance, dropout, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older,
2. possess a primary diagnosis of Tourette Syndrome or Persistent Tic Disorder,
3. fluent in English
4. residing in the United States,
5. either not be taking any tic suppressant medication or other psychotropic medication or be at a stable dose for 8 weeks prior to the baseline assessment and throughout the study

Exclusion Criteria:

1. be receiving concurrent psychotherapy for the duration of the study
2. have prior extensive experience with mindfulness and/or meditation and
3. cannot have another medical or psychological condition that would prevent the individual from fully engaging in the study or require a higher level of care (e.g., suicidality).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2018-08-07 (Actual); Study Completion 2018-08-07 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction Questionnaire | week 9

SECONDARY OUTCOMES:
Homework Compliance Questionnaire | Weeks 1-8
Attrition Form | Weeks 1-8
Adverse Events Monitoring Form | Weeks 1-9
Yale Global Tic Severity Scale (YGTSS) | Week 0, Week 9
Adult Tic Questionnaire | Weeks 0-9
Clinical Global Impressions Scale-Severity | Week 0, Week 9
Clinical Global Impressions Scale-Improvement | Week 9

OTHER OUTCOMES:
Yale-Brown Obsessive Compulsive Scale | Week 0, Week 9
Attention Deficit Hyperactivity Disorder Rating Scale | Week 0, Week 9
Patient Health Questionnaire-9 | Week 0, Week 9
Work and Social Adjustment Survey | Week 0, Week 9
Five Facet Mindfulness Questionnaire | Weeks 0-9
Credibility and Expectancy Questionnaire | Week 3
Self Compassion Scale | Week 0, Week 9
Affective Reactivity Index | Week 0, Week 9
Brief Irritability Test | Week 0, Week 9

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Reese, Ph.D., Principal Investigator — Bowdoin College
Locations (2):
- United States (2):
  - Bowdoin College, Brunswick, Maine
  - Massachusetts General Hospital, Boston, Massachusetts

REFERENCES:
- [Derived] Reese HE, Brown WA, Summers BJ, Shin J, Wheeler G, Wilhelm S. Feasibility and acceptability of an online mindfulness-based group intervention for adults with tic disorders. Pilot Feasibility Stud. 2021 Mar 24;7(1):82. doi: 10.1186/s40814-021-00818-y. PMID 33757602